CLINICAL TRIAL: NCT01748864
Title: A Single-Center Phase I Clinical Study to Evaluate The Biodistribution and Safety of 99mTC-Etarfolatide (EC20) in Normal Volunteers
Brief Title: Evaluation of the Biodistribution and Safety of 99mTC-Etarfolatide (EC20) in Normal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EC20.11
Record Dates: First submitted 2012-12-10; First posted 2012-12-13 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Volunteers

ARMS (1):
- Single Arm - Healthy Volunteers (Experimental): Etarfolatide (EC20)
  Interventions: Drug: Etarfolatide (EC20)

INTERVENTIONS:
Drug: Etarfolatide (EC20)

SUMMARY:
A Phase 1, single-center, open-label, single arm, baseline-controlled (for safety) study in normal volunteers. Study will determine biodistribution and excretion of the radioactive drug substance and evaluate the safety and tolerability of 99mTC-Etarfolatide in normal volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older.
* Subject must not have any major health problems as deemed by principal investigator.
* Subject must provide informed consent prior to enrollment.

Exclusion Criteria:

* Subject is pregnant or breast-feeding.
* Subject is simultaneously participating in another investigative drug or device study.
* Subject must have completed the follow-up phase of any previous study at least 30 days prior to enrollment in this study.
* Subject has a known history of chronic abuse of drugs or alcohol or tests positive in pre-study urine drug abuse screen.
* Subject is currently taking folic acid supplements and cannot stop taking the supplements for a period of 8 days (7 days prior to the study and one day after last imaging procedure).
* Subject's physical condition unsuitable for radionuclide imaging.
* Subject has been administered another radiopharmaceutical that would interfere with the assessment of the biodistribution of 99mTc-etarfolatide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Distribution of Radioactive Drug Substance | 24 hours
  To measure distribution of radioactivity from 99mTc-EC20 injection in blood and urine samples.

SECONDARY OUTCOMES:
Safety of 99mTc-Etarfolatide in Normal Volunteers | 4 days post-injection of EC20
  Asses any adverse events and serious adverse events experienced by volunteers.
Tolerability of 99mTc-Etarfolatide in Normal Volunteers | 4 days
  Asses any adverse events and serious adverse events experienced by volunteers.

OTHER OUTCOMES:
Quality of SPECT images of Normal Volunteers with or without injection of Folic Acid | 24 hours
  Comparison made of SPECT images taken of volunteers who received folic acid injection prior to 99mTc-EC20 injection and those who did not receive folic acid injection.
  Readability of scans, background "noise" as well as evaluation of any other differences will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Wael Harb, MD, Principal Investigator — Horizon Oncology Research, Inc.; Beth Safirstein, MD, Principal Investigator — MD Clinical
Locations (2):
- United States (2):
  - MD Clinical, Hallendale, Florida
  - Horizon Oncology, Lafayette, Indiana